CLINICAL TRIAL: NCT00127127
Title: A Phase I Clinical Study of L-001079038 in Patients With Solid Tumors
Brief Title: A Study of Vorinostat in Patients With Solid Tumors (MK-0683-029)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0683-029; 2005_040; MK-0683-029 (Other: Merck)
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Results first posted 2022-05-02 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Tumors
Keywords: Solid tumors
MeSH Terms: conditions — Neoplasms | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vorinostat 100 mg (Experimental): During Cycle 1, participants receive a single oral dose of vorinostat 100 mg on Day 1 in a fasted state, Day 3 in a fed state, and Day 19 in a fed state. On Days 5-18, participants receive vorinostat 100 mg twice daily, in the morning and evening. If participants do not match to the discontinuation criteria, they can continue the same dose level therapy during Cycle 2 and subsequent cycles. (Each cycle will be 26 days.)
  Interventions: Drug: vorinostat
- Vorinostat 200 mg (Experimental): During Cycle 1, participants receive a single oral dose of vorinostat 200 mg on Day 1 in a fasted state; on Day 3 in a fed state; and on Day 19 in a fed state. On Days 5-18, participants receive vorinostat 200 mg twice daily, in the morning and evening. If participants do not match to the discontinuation criteria, they can continue the same dose level therapy during Cycle 2 and subsequent cycles. (Each cycle will be 26 days.)
  Interventions: Drug: vorinostat
- Vorinostat 400 mg (Experimental): During Cycle 1, participants receive a single oral dose of vorinostat 400 mg on Day 1 in a fasted state; on Day 3 in a fed state; and on Day 19 in a fed state. On Days 5-18, participants receive a single oral dose of vorinostat 400 mg once-daily in the morning. If participants do not match to the discontinuation criteria, they can continue the same dose level therapy during Cycle 2 and subsequent cycles. (Each cycle will be 26 days.)
  Interventions: Drug: vorinostat
- Vorinostat 500 mg (Experimental): During Cycle 1, participants receive a single oral dose of vorinostat 500 mg on Day 1 in a fasted state; on Day 3 in a fed state; and on Day 19 in a fed state. On Days 5-18, participants receive a single oral dose of vorinostat 500 mg once-daily in the morning. If participants do not match to the discontinuation criteria, they can continue the same dose level therapy on the Cycle 2 and subsequent cycles.(Each cycle will be 26 days.)
  Interventions: Drug: vorinostat

INTERVENTIONS:
Drug: vorinostat — vorinostat 100 mg, 200 mg, 400 mg, or 500 mg single oral dose; once-daily or twice-daily administration
  Other Names: MK-0683; L-001079038; suberoylanilide hydroxamic acid (SAHA)

SUMMARY:
The primary purpose of this trial is to determine the maximum tolerated dose (MTD), or the maximum acceptable dose (MAD) and evaluate the dose limiting toxicity (DLT) of oral suberoylanilide hydroxamic acid in participants with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically or cytologically diagnosed solid tumor; no standard therapy available or participant has failed to respond to standard therapy

Exclusion Criteria:

* Participants with history of immunotherapy, radiotherapy, surgery, or chemotherapy during the previous 4 weeks; previous treatment is 5 or more chemotherapeutic regimens.
* Any uncontrolled concomitant illness
* Are pregnant or breast-feeding
* Serious drug or food allergy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-06-10 (Actual); Primary Completion 2009-08-21 (Actual); Study Completion 2009-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Fujiwara Y, Yamamoto N, Yamada Y, Yamada K, Otsuki T, Kanazu S, Iwasa T, Hardwick JS, Tamura T. Phase I and pharmacokinetic study of vorinostat (suberoylanilide hydroxamic acid) in Japanese patients with solid tumors. Cancer Sci. 2009 Sep;100(9):1728-34. doi: 10.1111/j.1349-7006.2009.01237.x. Epub 2009 May 31. PMID 19575752

RESULTS

PARTICIPANT FLOW:
Groups:
- Vorinostat 100 mg: During Cycle 1, participants received a single oral dose of vorinostat 100 mg on Day 1 (fasted), Day 3 (fed), and Day 19 (fed). On Days 5-18, participants received vorinostat 100 mg twice daily, in the morning and evening. If participants did not match to the discontinuation criteria, they could continue the same dose level therapy during Cycle 2 and subsequent cycles. (Each cycle was 26 days.)
- Vorinostat 200 mg: During Cycle 1, participants received a single oral dose of vorinostat 200 mg on Day 1 (fasted), Day 3 (fed), and Day 19 (fed). On Days 5-18, participants received vorinostat 200 mg twice daily, in the morning and evening. If participants did not match to the discontinuation criteria, they could continue the same dose level therapy during Cycle 2 and subsequent cycles. (Each cycle was 26 days.)
- Vorinostat 400 mg: During Cycle 1, participants received a single oral dose of vorinostat 400 mg on Day 1 (fasted), Day 3 (fed), Day 19 (fed). On Days 5-18, participants received a single oral dose of vorinostat 400 mg once-daily in the morning. If participants did not match to the discontinuation criteria, they could continue the same dose level therapy during Cycle 2 and subsequent cycles. (Each cycle was 26 days.)
- Vorinostat 500 mg: During Cycle 1, participants received a single oral dose of vorinostat 500 mg on Day 1 (fasted), Day 3 (fed), Day 19 (fed). On Days 5-18, participants received a single oral dose of vorinostat 500 mg once-daily in the morning. If participants did not match to the discontinuation criteria, they could continue the same dose level therapy on the Cycle 2 and subsequent cycles.(Each cycle was 26 days.)
Period: Overall Study
Arm/Group | Vorinostat 100 mg | Vorinostat 200 mg | Vorinostat 400 mg | Vorinostat 500 mg
Started | 3 | 6 | 3 | 6
Completed | 2 | 1 | 3 | 3
Not Completed | 1 | 5 | 0 | 3
Not completed — Adverse Event | 0 | 2 | 0 | 1
Not completed — Lack of Efficacy | 1 | 3 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vorinostat 100 mg | Vorinostat 200 mg | Vorinostat 400 mg | Vorinostat 500 mg | Total
Number analyzed (Participants) | 3 | 6 | 3 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.7 (6.7) | 60.5 (6.3) | 49.3 (21.5) | 57.7 (8.3) | 57.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 0 | 0 | 3
  Male | 3 | 3 | 3 | 6 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 6 | 3 | 6 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced One or More Adverse Events
Description: An adverse event is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to approximately 4 years
Population: All participants who received at least one dose of study drug. (Note: 1 participant in 200 mg treatment group had dose reduced to 100 mg in Cycle 8 and is also included in 100 mg treatment group for adverse events.)
Measure: Count of Participants; unit: Participants
Groups:
- Vorinostat 500 mg: During Cycle 1, participants received a single oral dose of vorinostat 500 mg on Day 1 (fasted), Day 3 (fed), Day 19 (fed). On Days 5-18, participants received a single oral dose of vorinostat 500 mg once-daily in the morning. If participants did not match to the discontinuation criteria, they could continue the same dose level therapy on the Cycle 2 and subsequent cycles. (Each cycle was 26 days.)
Arm/Group | Vorinostat 100 mg | Vorinostat 200 mg | Vorinostat 400 mg | Vorinostat 500 mg
Number analyzed (Participants) | 4 | 6 | 3 | 6
Participants | 4 | 6 | 3 | 6

2. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event
Description: as for outcome 1
Time Frame: Up to approximately 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vorinostat 100 mg | Vorinostat 200 mg | Vorinostat 400 mg | Vorinostat 500 mg
Number analyzed (Participants) | 4 | 6 | 3 | 6
Participants | 0 | 1 | 0 | 1

3. Primary Outcome: Number of Participants With a Dose-Limiting Toxicity (DLT) During Cycle 1
Description: A DLT was defined as an event considered to be related to study treatment and included: 1) Grade 4 neutropenia refractory to treatments persisting more than 5 days; 2) Grade 3 or more severe neutropenic fever; 3) Grade 3 thrombocytopenia requiring blood transfusions or Grade 4 thrombocytopenia; 4) Grade 4 hemoglobin decrease; 5) Grade 3 or more severe non-hematological toxicities other than anorexia, nausea/vomiting, and fatigue. (For the diarrhea, it was defined as not to use the frequency for the grading. For the alanine aminotransferase [ALT]/aspartate aminotransferase [AST]), it was defined as the case of over 300 IU/L; 6) Grade 3 or more severe anorexia, nausea/vomiting, and fatigue refractory to treatments; and 7) compliance of the study drug, while administrating 14 consecutive days, was less than 50% due to the drug-related adverse experience.
Time Frame: Up to 26 days
Population: All participants who received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Groups:
- Vorinostat 100 mg: During Cycle 1, participants received a single oral dose of vorinostat 100 mg on Day 1 (fasted), Day 3 (fed), and Day 19 (fed). On Days 5-18, participants received vorinostat 100 mg twice daily, in the morning and evening. (Cycle 1 was 26 days.)
- Vorinostat 200 mg: During Cycle 1, participants received a single oral dose of vorinostat 200 mg on Day 1 (fasted), Day 3 (fed), and Day 19 (fed). On Days 5-18, participants received vorinostat 200 mg twice daily, in the morning and evening. (Cycle 1 was 26 days.)
- Vorinostat 400 mg: During Cycle 1, participants received a single oral dose of vorinostat 400 mg on Day 1 (fasted), Day 3 (fed), Day 19 (fed). On Days 5-18, participants received a single oral dose of vorinostat 400 mg once-daily in the morning. (Cycle 1 was 26 days.)
- Vorinostat 500 mg: During Cycle 1, participants received a single oral dose of vorinostat 500 mg on Day 1 (fasted), Day 3 (fed), Day 19 (fed). On Days 5-18, participants received a single oral dose of vorinostat 500 mg once-daily in the morning. (Cycle 1 was 26 days.)
Arm/Group | Vorinostat 100 mg | Vorinostat 200 mg | Vorinostat 400 mg | Vorinostat 500 mg
Number analyzed (Participants) | 3 | 6 | 3 | 6
Participants | 0 | 3 | 0 | 2

4. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Hour 0 to Infinity (AUC0-inf) of Vorinostat After a Single Oral Dose in a Fasted State
Description: AUC0-inf is the area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time.
Time Frame: Day 1: pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours post-dose
Population: All participants who complied with the protocol and had Day 1 pharmacokinetic (PK) data for AUC0-inf.
Measure: Geometric Mean (Standard Deviation); unit: μM·hours
Groups:
- Vorinostat 100 mg FASTED: Participants received a single oral dose of vorinostat 100 mg in fasted state on Day 1.
- Vorinostat 200 mg FASTED: Participants received a single oral dose of vorinostat 200 mg in fasted state on Day 1.
- Vorinostat 400 mg FASTED: Participants received a single oral dose of vorinostat 400 mg in fasted state on Day 1.
- Vorinostat 500 mg FASTED: Participants received a single oral dose of vorinostat 500 mg in fasted state on Day 1.
Arm/Group | Vorinostat 100 mg FASTED | Vorinostat 200 mg FASTED | Vorinostat 400 mg FASTED | Vorinostat 500 mg FASTED
Number analyzed (Participants) | 3 | 6 | 3 | 6
μM·hours | 1.20 (0.27) | 2.31 (0.96) | 3.96 (1.62) | 3.47 (2.21)

5. Secondary Outcome: AUC0-Inf of Vorinostat After a Single Oral Dose in a Fed State
Description: as for outcome 4
Time Frame: Day 3: pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours post-dose
Population: All participants who complied with the protocol and had Day 3 PK data for AUC0-inf.
Measure: Geometric Mean (Standard Deviation); unit: μM·hours
Groups:
- Vorinostat 100 mg FED: Participants received a single oral dose of vorinostat 100 mg in a fed state on Day 3.
- Vorinostat 200 mg FED: Participants received a single oral dose of vorinostat 200 mg in a fed state on Day 3.
- Vorinostat 400 mg FED: Participants received a single oral dose of vorinostat 400 mg in a fed state on Day 3.
- Vorinostat 500 mg FED: Participants received a single oral dose of vorinostat 500 mg in a fed state on Day 3.
Arm/Group | Vorinostat 100 mg FED | Vorinostat 200 mg FED | Vorinostat 400 mg FED | Vorinostat 500 mg FED
Number analyzed (Participants) | 3 | 6 | 3 | 6
μM·hours | 0.98 (0.07) | 2.22 (0.89) | 4.30 (0.37) | 5.93 (1.78)

6. Secondary Outcome: AUC0-inf of Vorinostat After 14 Days of Once-Daily or Twice-Daily Administration
Description: as for outcome 4
Time Frame: Day 19: pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours post-dose
Population: All participants who complied with the protocol and had up to Day 19 PK data for AUC0-inf
Measure: Geometric Mean (Standard Deviation); unit: μM·hours
Groups:
- Vorinostat 100 mg Twice-daily: Participants received Vorinostat 100 mg twice daily, in the morning and evening, for 14 days (Days 5-18).
- Vorinostat 200 mg Twice-daily: Participants received vorinostat 200 mg twice daily, in the morning and evening, for 14 days (Days 5-18).
- Vorinostat 400 mg Once-daily: Participants received vorinostat 400 mg once daily in the morning for 14 days (Days 5-18).
- Vorinostat 500 mg Once-daily: Participants received vorinostat 500 mg once daily in the morning for 14 days (Days 5-18).
Arm/Group | Vorinostat 100 mg Twice-daily | Vorinostat 200 mg Twice-daily | Vorinostat 400 mg Once-daily | Vorinostat 500 mg Once-daily
Number analyzed (Participants) | 3 | 5 | 3 | 5
μM·hours | 1.33 (0.23) | 2.76 (0.85) | 5.41 (2.18) | 6.33 (1.53)

7. Secondary Outcome: Maximum Concentration (Cmax) of Vorinostat After a Single Oral Dose in a Fasted State
Description: Cmax is a measure of the maximum amount of drug in the plasma after the dose is given.
Time Frame: Day 1: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours post-dose
Population: All participants who complied with the protocol and had Day 1 PK data for Cmax
Measure: Geometric Mean (Standard Deviation); unit: μM
Groups:
- Vorinostat 200 mg FASTED: Participants received single oral dose of vorinostat 200 mg on Day 1 in a fasted state.
- Vorinostat 400 mg FASTED: Participants received a single oral dose of vorinostat 400 mg on Day 1 in a fasted state.
- Vorinostat 500 mg FASTED: Participants received a single oral dose of vorinostat 500 mg on Day 1 in a fasted state.
Arm/Group | Vorinostat 100 mg FASTED | Vorinostat 200 mg FASTED | Vorinostat 400 mg FASTED | Vorinostat 500 mg FASTED
Number analyzed (Participants) | 3 | 6 | 3 | 6
μM | 0.49 (0.15) | 0.77 (0.13) | 1.19 (0.20) | 1.06 (0.52)

8. Secondary Outcome: Cmax of Vorinostat After a Single Oral Dose in a Fed State
Description: Cmax is a measure of the maximum amount of drug in the plasma after the dose is given.
Time Frame: Day 3: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours post-dose
Population: All participants who complied with the protocol and had Day 3 PK data for Cmax
Measure: Geometric Mean (Standard Deviation); unit: μM
Arm/Group | Vorinostat 100 mg FED | Vorinostat 200 mg FED | Vorinostat 400 mg FED | Vorinostat 500 mg FED
Number analyzed (Participants) | 3 | 6 | 3 | 6
μM | 0.21 (0.14) | 0.59 (0.22) | 0.93 (0.12) | 1.35 (0.39)

9. Secondary Outcome: Cmax of Vorinostat After 14 Days of Once-Daily or Twice-Daily Administration
Description: Cmax is a measure of the maximum amount of drug in the plasma after the dose is given.
Time Frame: Day 19: pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours post-dose
Population: All participants who complied with the protocol and had up to Day 19 PK data for Cmax
Measure: Geometric Mean (Standard Deviation); unit: μM
Arm/Group | Vorinostat 100 mg Twice-daily | Vorinostat 200 mg Twice-daily | Vorinostat 400 mg Once-daily | Vorinostat 500 mg Once-daily
Number analyzed (Participants) | 3 | 5 | 3 | 5
μM | 0.29 (0.25) | 0.84 (0.56) | 0.86 (0.61) | 1.09 (0.30)

10. Secondary Outcome: Time to Maximum Concentration (Tmax) of Vorinostat After a Single Oral Dose in a Fasted State
Description: Tmax is a measure of the time to reach the maximum concentration in the plasma after the drug dose.
Time Frame: Day 1: pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours post-dose
Population: All participants who complied with the protocol and had Day 1 PK data for Tmax
Measure: Mean (Standard Deviation); unit: Hours
Groups:
- Vorinostat 100 mg FASTED: Participants received a single oral dose of vorinostat 100 mg in a fasted state on Day 1.
- Vorinostat 200 mg FASTED: Participants received a single oral dose of vorinostat 200 mg in a fasted state on Day 1.
- Vorinostat 400 mg FASTED: Participants received a single oral dose of vorinostat 400 mg in a fasted state on Day 1.
- Vorinostat 500 mg FASTED: Participants received a single oral dose of vorinostat 500 mg in a fasted state on Day 1.
Arm/Group | Vorinostat 100 mg FASTED | Vorinostat 200 mg FASTED | Vorinostat 400 mg FASTED | Vorinostat 500 mg FASTED
Number analyzed (Participants) | 3 | 6 | 3 | 6
Hours | 0.84 (0.30) | 1.59 (0.74) | 2.49 (0.86) | 1.91 (0.91)

11. Secondary Outcome: Tmax of Vorinostat After a Single Oral Dose in a Fed State
Description: Tmax is a measure of the time to reach the maximum concentration in the plasma after the drug dose.
Time Frame: Day 3: pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours post-dose
Population: All participants who complied with the protocol and had Day 3 PK data for Tmax
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Vorinostat 100 mg FED | Vorinostat 200 mg FED | Vorinostat 400 mg FED | Vorinostat 500 mg FED
Number analyzed (Participants) | 3 | 6 | 3 | 6
Hours | 5.66 (3.79) | 3.00 (0.89) | 3.53 (2.33) | 3.17 (1.17)

12. Secondary Outcome: Tmax of Vorinostat After 14 Days of Once-Daily or Twice-Daily Administration
Description: Tmax is a measure of the time to reach the maximum concentration in the plasma after the drug dose.
Time Frame: Day 19: pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours post-dose
Population: All participants who complied with the protocol and had up to Day 19 PK data for Tmax
Measure: Mean (Standard Deviation); unit: Hours
Groups:
- Vorinostat 400 mg Once-daily: Participants received vorinostat 400 mg once daily for 14 days (Days 5-18).
- Vorinostat 500 mg Once-daily: Participants received vorinostat 500 mg once daily for 14 days (Days 5-18).
Arm/Group | Vorinostat 100 mg Twice-daily | Vorinostat 200 mg Twice-daily | Vorinostat 400 mg Once-daily | Vorinostat 500 mg Once-daily
Number analyzed (Participants) | 3 | 5 | 3 | 5
Hours | 4.66 (1.16) | 3.30 (1.10) | 4.34 (1.53) | 4.61 (1.95)

13. Secondary Outcome: Apparent Terminal Half-Life (t½) of Vorinostat After a Single Oral Dose in a Fasted State
Description: t½ is the elimination half-life of study drug. t½ is the time it takes for half of the study drug in the blood plasma to dissipate.
Time Frame: Day 1: pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours post-dose
Population: All participants who complied with the protocol and had Day 1 PK data for t½
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Vorinostat 100 mg FASTED | Vorinostat 200 mg FASTED | Vorinostat 400 mg FASTED | Vorinostat 500 mg FASTED
Number analyzed (Participants) | 3 | 6 | 3 | 6
Hours | 1.08 (0.30) | 1.83 (0.53) | 1.90 (0.72) | 1.93 (0.67)

14. Secondary Outcome: t½ of Vorinostat After a Single Oral Dose in a Fed State
Description: as for outcome 13
Time Frame: Day 3: pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours post-dose
Population: All participants who complied with the protocol and had Day 3 PK data for t½
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Vorinostat 100 mg FED | Vorinostat 200 mg FED | Vorinostat 400 mg FED | Vorinostat 500 mg FED
Number analyzed (Participants) | 2 | 6 | 3 | 6
Hours | 1.62 (0.45) | 1.36 (0.28) | 2.01 (1.47) | 1.60 (0.66)

15. Secondary Outcome: t½ of Vorinostat After 14 Days of Once-Daily or Twice-Daily Administration
Description: as for outcome 13
Time Frame: Day 19: pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours post-dose
Population: All participants who complied with the protocol and had up to Day 19 PK data for t½
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Vorinostat 100 mg Twice-daily | Vorinostat 200 mg Twice-daily | Vorinostat 400 mg Once-daily | Vorinostat 500 mg Once-daily
Number analyzed (Participants) | 3 | 5 | 2 | 5
Hours | 1.95 (0.54) | 1.42 (0.50) | 1.98 (1.56) | 1.30 (0.41)

ADVERSE EVENTS:
Time Frame: Up to approximately 4 years
Description: Serious Adverse Events and Other Adverse Events: All participants who received at least one dose of study treatment. All-Cause Mortality: All participants included in a treatment group at enrollment, regardless of treatment duration. (Note: 1 participant in 200 mg treatment group had dose reduced to 100 mg in Cycle 8 and is also included in 100 mg treatment group for adverse events.)
Arm/Group | Vorinostat 100 mg | Vorinostat 200 mg | Vorinostat 400 mg | Vorinostat 500 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/6 | 1/3 | 0/6
Other Adverse Events (participants affected / at risk) | 4/4 | 6/6 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat 100 mg (N=4) | Vorinostat 200 mg (N=6) | Vorinostat 400 mg (N=3) | Vorinostat 500 mg (N=6)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat 100 mg (N=4) | Vorinostat 200 mg (N=6) | Vorinostat 400 mg (N=3) | Vorinostat 500 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 5 (12) | 1 (3) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 5 (17) | 2 (2) | 4 (7)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (6) | 2 (3) | 1 (4)
Chest discomfort (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 5 (17) | 2 (3) | 5 (9)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (13) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (5) | 0 (0) | 1 (1)
Blood albumin decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 3 (12) | 0 (0) | 2 (3)
Blood calcium decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood chloride decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Blood cholesterol decreased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 2 (11) | 0 (0) | 0 (0)
Blood creatine phosphokinase MB increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (2) | 3 (14) | 0 (0) | 1 (2)
Blood glucose increased (Investigations) | 1 (3) | 2 (2) | 1 (2) | 4 (7)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 2 (17) | 0 (0) | 1 (1)
Blood magnesium increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Blood sodium decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Blood triglycerides decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blood uric acid decreased (Investigations) | 0 (0) | 2 (4) | 0 (0) | 1 (1)
Electrocardiogram ST-T change (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Glucose urine present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 3 (6) | 0 (0) | 1 (2)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 2 (3)
Neutrophil count decreased (Investigations) | 2 (6) | 5 (60) | 0 (0) | 1 (2)
Platelet count decreased (Investigations) | 1 (2) | 6 (35) | 3 (5) | 4 (9)
Protein total decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 3 (4) | 0 (0) | 1 (1)
Red blood cell count decreased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 2 (6) | 1 (9) | 1 (1) | 2 (2)
White blood cell count decreased (Investigations) | 1 (3) | 5 (30) | 0 (0) | 1 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 3 (11) | 2 (4) | 5 (12)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heat rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.